CLINICAL TRIAL: NCT03662581
Title: Evaluating a Primary-Care Group-based Mindfulness Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 caused the program to change in its delivery to virtual, therefore it no longer followed the intervention described in the protocol.
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Elizabeth Alvarez, Assistant Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Group-based Mindfulness
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Anxiety; Depression; Sleep Initiation and Maintenance Disorders; Social Isolation
Keywords: Generalized anxiety disorder; Mental health; Mindfulness; Group-based therapy
MeSH Terms: conditions — Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders; Social Isolation; Generalized Anxiety Disorder; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study evaluates the effect of the intervention using a single group, before-after study model. The subjects will be evaluated at baseline and followed longitudinally, until study completion and a long-term followup.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Group Program (Experimental): A primary care mindfulness-based rolling admissions program where subjects must attend 4 of 8 consecutive group sessions, to be considered to have completed the program.
  Interventions: Behavioral: Mindfulness Group Program

INTERVENTIONS:
Behavioral: Mindfulness Group Program — The mindfulness program has the following aims (Iacono, 2018): to teach mindfulness skills for stress reduction, self-compassion, and dealing with difficult thoughts and emotions, to promote an integrative concept of health, which treats the whole person, to promote community building and positive relationships, and to capitalize on the power of groups to:
  1. Foster peer-to-peer learning and support when it comes to coping with life challenges
  2. Combat isolation
  3. Increase efficiency, quality, and timeliness of care

SUMMARY:
The study evaluates the effectiveness of a group-based mindfulness program conducted in a primary care setting. This study also aims to identify any scale-up and implementation considerations for the program.

DETAILED DESCRIPTION:
A primary care group-based mindfulness program was developed by community physicians and co-op and public health students in Ajax, Ontario. The program was started in January 2018 and is run through the Ajax Harwood Clinic, which is a clinic housing a Family Health Organization (FHO) comprising of 5 physicians and approximately 6,500 patients. The purposes of the program are:

1. To teach mindfulness skills for stress reduction, self-compassion, and dealing with difficult thoughts and emotions,
2. To promote an integrative concept of health, which treats the whole person
3. To promote community building and positive relationships
4. To capitalize on the power of groups to:

   1. Foster peer-to-peer learning and support when it comes to coping with life challenges
   2. Combat isolation
   3. Increase efficiency, quality, and timeliness of care

This study evaluates the 8-week rolling admission mindfulness program, by first doing a retrospective chart review to identify effect sizes and then conducting a before-after study evaluation of the effect of the mindfulness program on key mental health outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled in mindfulness-based program through Ajax Harwood Clinic
* Age of 18
* English-speaking ability to participate in program
* Able to provide informed consent

Exclusion Criteria:

* no formal exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder - 7 (GAD-7) | Change from baseline each week until 8 weeks and at 8 months post-baseline
  The GAD-7 is a validated instrument for the diagnosis and treatment response of anxiety disorders (Spitzer et al, 2006; Hinz et al, 2017). It is comprised of 7 questions with 4 answer options, ranging from "not at all" to "nearly every day" and scored 0-3 with a total score ranging from 0-21 (Spitzer et al, 2006). Scores of 5-9, 10-14, and 15-21 represent mild, moderate and severe generalized anxiety disorder, respectively. In the primary care setting, the GAD-7 has high diagnostic validity, with a threshold of 10 exhibiting a sensitivity of 89% and specificity of 82% for generalized anxiety disorder (Spitzer et al, 2006). Other conditions related to generalized anxiety disorder including panic disorder, social anxiety disorder and post-traumatic stress disorder have also been sensitive to a GAD-7 score of 10 (Kroenke et al, 2007).

SECONDARY OUTCOMES:
Patient Heath Questionnaire 9 (PHQ-9) for depression | Change from baseline each week until 8 weeks and at 8 months post-baseline
  The Patient Health Questionnaire-9 (PHQ-9) is made up of nine questions and is diagnostic for depression. Importantly, the PHQ-9 has also been found to be sensitive to change for monitoring of treatment outcomes (Kohrt et al, 2016; Lowe et al, 2004). The PHQ-9 asks participants, "Over the last 2 weeks, how often have you been bothered by any of the following problems?" All answers have four options ranging from "not at all," "several days," more than half the days," or "nearly every day" for a number of symptoms related to depression. Major depression and other depressive syndromes are diagnosed based on answers of "more than half the days" or "nearly every day" to "Little interest or pleasure in doing things" or "Feeling down, depressed, or hopeless" plus 2-5 or more of the other symptoms.
Insomnia Severity Index (ISI) | Change from baseline each week until 8 weeks and at 8 months post-baseline
  The Insomnia Severity Index, a 7-item scale, was identified as the most fitting validated scale to identify insomnia symptoms (Bastien et al., 2001). Each of the questions is measured on a scale of 0-4 and the answers are added up to get a total score.
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
DeJong Gierveld Loneliness Scale | Change from baseline each week until 8 weeks and at 8 months post-baseline
  The DeJong Gierveld 6-item Loneliness Scale captures both emotional loneliness (missing an intimate relationship) and social loneliness (missing a wider social network) (Gierveld et al, 2006; Grygiel et al, 2016). Each subscale is made up of three questions with possible answers of "yes," "more or less," or "no." Questions 1-3 are negatively worded and answers of "yes" or "more or less" are scored as "1", while "no" is scored as "0". On positively worded questions (4-6), neutral or negative answers ("no" or "more or less") are scored as "1," while "yes" is scored as "0." This gives a range of 0 (not lonely)-3 (very lonely) in each subscale, or 0 (not lonely)-6 (very lonely) in the total scale. However, we have changed this scoring so that we can further discriminate between neutral and other answers. Therefore, our scoring on each question ranges from 0-2, giving a total scale of 0 (not lonely)-12 (very lonely).

OTHER OUTCOMES:
Hemoglobin A1C (HgA1C) | Change from baseline at 8 weeks and at 8 months post-baseline
  Assessing prevalence of diabetes via HgA1C levels from electronic medical record (EMR) for comorbidity comparison
Weight | Change from baseline at 8 weeks and at 8 months post-baseline
  Assessing prevalence of obesity/comorbidities from weight through EMR data

CONTACTS AND LOCATIONS:
Overall Officials: Yaswanta Gummadi, BHSc, Principal Investigator — McMaster University; Elizabeth Alvarez, MD, Principal Investigator — McMaster University
Locations (1):
- Ajax Harwood Clinic, Ajax, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Hinz A, Klein AM, Brahler E, Glaesmer H, Luck T, Riedel-Heller SG, Wirkner K, Hilbert A. Psychometric evaluation of the Generalized Anxiety Disorder Screener GAD-7, based on a large German general population sample. J Affect Disord. 2017 Mar 1;210:338-344. doi: 10.1016/j.jad.2016.12.012. Epub 2016 Dec 18. PMID 28088111
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Kohrt BA, Luitel NP, Acharya P, Jordans MJ. Detection of depression in low resource settings: validation of the Patient Health Questionnaire (PHQ-9) and cultural concepts of distress in Nepal. BMC Psychiatry. 2016 Mar 8;16:58. doi: 10.1186/s12888-016-0768-y. PMID 26951403
- [Background] Lowe B, Unutzer J, Callahan CM, Perkins AJ, Kroenke K. Monitoring depression treatment outcomes with the patient health questionnaire-9. Med Care. 2004 Dec;42(12):1194-201. doi: 10.1097/00005650-200412000-00006. PMID 15550799
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Gierveld, J. D. J., & Tilburg, T. V. (2006). A 6-Item Scale for Overall, Emotional, and Social Loneliness: Confirmatory Tests on Survey Data. Research on Aging, 28(5), 582-598. https://doi.org/10.1177/0164027506289723
- [Background] Grygiel P, Humenny G, Rebisz S. Using the De Jong Gierveld Loneliness Scale With Early Adolescents: Factor Structure, Reliability, Stability, and External Validity. Assessment. 2019 Mar;26(2):151-165. doi: 10.1177/1073191116682298. Epub 2016 Dec 8. PMID 27932403